CLINICAL TRIAL: NCT00176241
Title: A Phase I Trial of Biweekly Gemcitabine & Paclitaxel & Low-Dose Fractionated Radiation in the Treatment of Metastatic or Recurrent Head & Neck Cancer
Brief Title: Phase I Trial of Biweekly Gemcitabine & Paclitaxel & Low-Dose Radiation for Metastatic or Recurrent Head & Neck Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Susanne Arnold (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor-Investigator, Susanne Arnold, Principal Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-H&N-16-EL
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Head and Neck Cancer
Keywords: head and neck; Gemcitabine; Paclitaxel; radiation; low-dose radiation; recurrent; metastatic
MeSH Terms: conditions — Head and Neck Neoplasms; Recurrence; Neoplasm Metastasis | interventions — Gemcitabine; Paclitaxel; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: gemcitabine; Drug: paclitaxel; Radiation: radiation

INTERVENTIONS:
Drug: gemcitabine — 2000-3000mg/m2 IV on days 1 & 15
  Other Names: Gemzar
Drug: paclitaxel — 150 mg/m2 IV on days 1 & 15
Radiation: radiation — 50-80 cGy on days 1,2,15,16

SUMMARY:
This study seeks to establish the safety of gemcitabine, paclitaxel and low-dose radiation in recurrent, metastatic head and neck cancer through a two-stage dose escalation study, first with Gemcitabine dose escalation and then with low-dose radiation escalation.

Treatment Schedule

Treatment will be administered on an inpatient or outpatient basis.

* Gemcitabine:2000 to 3000mg/m2 IV (in the vein) on days 1 and 15 every 28 days over 30-60 minutes.
* Paclitaxel: 150 mg/m2 IV(in the vein)on days 1 and 15 every 28 days over 60 minutes.
* Low Dose Radiation: 50-80 cGy twice daily on days 1, 2, 15, & 16 every 28 days at least 4 hours apart.

DETAILED DESCRIPTION:
Objectives:

1. To assess the MTD of low-dose fractionated radiation in combination with Gemcitabine and Paclitaxel in recurrent or metastatic head and neck cancer in the relapsed setting.

Secondary Objectives:

1. To assess quantitative toxicities in this group of patients treated with this regimen.
2. To assess response rate in this group of patients treated with this regimen
3. To investigate in an exploratory manner, the association of tumor markers p53, p21waf1/cip1, bcl-xL, bcl-2 and bax (evaluated by immunohistochemistry) with response rate using pre- and post-treatment biopsies.

This study seeks to establish the safety of gemcitabine, paclitaxel and low-dose radiation in recurrent, metastatic head and neck cancer through a two-stage dose escalation study, first with Gemcitabine dose escalation and then with low-dose radiation escalation.

Treatment Schedule:

Treatment will be administered on an inpatient or outpatient basis.

* Gemcitabine:2000 to 3000mg/m2 IV on days 1 and 15 every 28 days over 30-60 minutes.
* Paclitaxel: 150 mg/m2 IV on days 1 and 15 every 28 days over 60 minutes.
* Low Dose Radiation: 50-80 cGy twice daily on days 1, 2, 15, & 16 every 28 days at least 4 hours apart.

ELIGIBILITY:
Inclusion Criteria:

1. 18 yrs old or greater & have histologically or cytologically proven metastatic or recurrent head & neck cancer & have failed at least 1 prior, but not more than 3 chemotherapeutic regimen. Patients who have recurred after previous surgery and/or radiation may participate in this trial, & patients may have had prior neoadjuvant or adjuvant therapy. No restriction is placed on the # of cycles (beyond 1) of prior therapy, however, patients must not have received the combination of Gemcitabine & Paclitaxel previously.
2. Patients with known brain metastases are eligible for this trial if disease has been treated & the patient is clinically stable & documented by a stable or improved pretreatment CT or MRI of the brain to evaluate CNS disease within 28 days prior to registration.
3. Patients must have measurable OR non-measurable disease documented by CT, MRI, X-ray or nuclear exam (FDG-PET). Measurable disease must be assessed within 28 days prior to registration & non-measurable must be assessed within 42 days prior to registration. Pleural effusions, ascites & lab parameters are not acceptable as only evidence of disease.
4. Patients must have progressed after at least 1 prior chemotherapeutic regimen. Prior biologic therapy or radiation is permitted; however, at least 2 wks must have elapsed since completion of prior therapy & patients must have recovered from all associated toxicities at time of registration.
5. At least 3 wks must have elapsed since surgery (thoracic or other major surgeries) & patients must have recovered from all associated toxicities at time of registration. Measurable or non-measurable disease must be present outside the area of surgical resection.
6. Patients must have an ANC 1,500/µl & platelet count 100,000/µl obtained within 28 days prior to registration.
7. Patients must have adequate hepatic function documented by a serum bilirubin 1.5 x institutional ULN & LFTs (SGOT or SGPT) 2.5 x the institutional ULN obtained within 28 days prior to registration.
8. All patients with pulmonary metastasis must have an FEV1 of > 1000 ml/min obtained within 28 days prior to registration & must have PFTs with DLCO.
9. All patients must have a Zubrod Performance Status of 0,1 or 2.
10. Peripheral neuropathy, if present, must be Grade 1.
11. Patients must be informed of investigational nature of this study & must sign & give written informed consent in accordance with institutional & federal guidelines.

Exclusion Criteria:

1. No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated Stage I or II cancer from which the patient is currently in complete remission or other cancer from which the patient has been disease-free for 5 yrs.
2. Pregnant or nursing women may not participate in this trial because of the increased risk of fetal harm including fetal death from the chemotherapeutic agents. Women/men of reproductive potential may not participate unless they have agreed to use an effective contraceptive method (hormonal or barrier method of birth control; abstinence) prior to study entry & for duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
3. Patients taking drugs that are strong inducers of the enzyme CYP3A4 including anticonvulsants (i.e., phenytoin, phenobarbital, carbamazepine, or primidone) & rifampin OR strong inhibitors of CYP3A4 (clarithromycin, itraconazole, and ketoconazole) will be excluded from this study. Patients must be off these medications for 2 wks in order to participate in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2005-12; Primary Completion 2008-09 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | toxicity notations made during weeks 3, 5, 7 & 9 of each cycle

SECONDARY OUTCOMES:
Toxicity | weeks 3, 5, 7 & 9 of each cycle & also evaluated throughout study by weekly CBC
Response rate | assessed pre-study & week 8 and as needed during follow-up.
Association of tumor markers p53, p21waf1/cip1, bcl-xL, bcl-2 & bax with response rate | patients who consent to biopsy, obtain pre-study & 3-24 hrs after completion of 4th fraction of radiation, evaluated by immunohistochemistry

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Arnold, MD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

REFERENCES:
- See also: Markey Cancer Center clinical trials search — http://markey.uky.edu/studysearch/default.aspx